CLINICAL TRIAL: NCT03430934
Title: Near Infra-Red Navigation (NAVI) System for Mohs Tumor Mapping
Brief Title: Non-invasive Fluorescent Imaging System for Imaging Mohs Tumor
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Nicholas J Golda, Clinical Associate Professor, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2009753
Record Dates: First submitted 2018-02-06; First posted 2018-02-13 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Skin Cancer
Keywords: Mohs tumor
MeSH Terms: conditions — Skin Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Intervention Model Description: Evaluation of a in-house developed Near Infrared Navigation System camera for Moh's tumor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- NAVI mapping with Indocyanine green (Experimental): Participants will undergo their scheduled Mohs surgery with the addition of the NAVI mapping with ICG dye
  Interventions: Combination Product: NAVI mapping with Indocyanine green

INTERVENTIONS:
Combination Product: NAVI mapping with Indocyanine green — Moh's tumor imaging with Indocyanine green
  Other Names: Imaging of skin tumor; Indocyanine green

SUMMARY:
The objective of this study is to correlate traditional histological Mohs tissue mapping of a cutaneous tumor with the ICG-mapping procedure. The use of intradermal ICG in a cutaneous tumor during MMS followed by visualization using a fluorescent imaging system could allow surgeons to directly visualize, and roughly map the extent of a primary skin cancer and plan the Mohs procedure (i.e. the initial excision size and subsequent layer widths) accordingly.

DETAILED DESCRIPTION:
The incidence of non-melanoma skin cancers, i.e. basal cell and squamous cell carcinoma (BCC and SCC), in the US is over 5.4 million. Of these, BCC represents the majority, with an incidence of over 4 million. Recent guidelines published on the treatment of BCC and SCC establish Mohs micrographic surgery (MMS) as the treatment of choice for high-risk SCCs and BCCs and for those in cosmetically sensitive locations.

MMS involves the step-wise removal and subsequent histological examination of thin layers of cancer containing skin until only cancer-free tissue remains. At the initial layer, only clinically involved skin is excised. The excised tumor is oriented using purposeful marks on the tissue and color-coding. Using this orientation, a "Mohs map" is drawn to indicate where malignancy is seen histologically. For each following layer, orientation is maintained, and only margins with remaining malignant tissue are removed as indicated on the map. As the goal is to spare as much normal tissue as possible, Mohs layers are only a few millimeters thin. The average number of layers needed to remove an entire tumor per Mohs case is cited as 1.74. However, outlier providers - that take a fewer or higher number of layers to clear a cancer- do exist. While this could represent providers who see more complicated cases, and skin tumors are often more extensive than initially clinically apparent, the need to balance efficiency with the width of a layer likely also plays a role.

Fluorescence image guided surgery using Indocyanine green (ICG), an FDA approved near-infrared (NIR) dye, has been used for effective visualization of intra-osseous tumoral tissues in real-time, allowing surgeons to make intraoperative decisions for further resection of otherwise clinically-uninvolved tissue. The use of intradermal ICG in a cutaneous tumor during MMS could allow surgeons to directly visualize, and roughly map the extent of a primary skin cancer preoperatively and plan the Mohs procedure (i.e. the initial excision size and subsequent layer widths) accordingly. No current such mapping system exists for use in cutaneous tumors.

Thus, while MMS represents an effective methodology to remove malignant tissue and spare as much normal skin as possible, it is a lengthy process totaling several hours, and given the need for histological processing at each stage, its duration primarily correlates with the number of layers or stages needed. A pre-operative map of the extent of the tumor could allow for: (1) a larger first layer - on the initial excision, only clinically evident tumor is excised, but skin tumors are at times more extensive that clinically apparent; and the Mohs surgeon to take thicker subsequent layers as needed. Effective and accurate pre-operative tumor mapping with ICG therefore has the potential to reduce the total number of Mohs layers taken for a patient. This is effect would improve patient safety and quality of care, and reduce unnecessary financial burden associated with outliers. As a decreased number of layers would directly shorten the total procedure length, preoperative mapping also has the potential to help increase patient access to MMS.

ELIGIBILITY:
Inclusion Criteria:

Subjects who are scheduled to undergo Mohs surgery for a basal cell carcinoma tumor, with a minimum tumor size of 1.5 cm, will be selected for the study procedure. A total of 10 subjects are required to complete the study. We will need to consent 15 subjects to achieve a total of 10 subjects to complete the study.

* Individuals 18 years or older
* All races and ethnicity
* Smokers and non-smokers

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Near Infra-Red Navigation (NAVI) System for Mohs Tumor Mapping | 24 HOURS
  Correlation of traditional histological Mohs tissue mapping of a cutaneous tumor with the ICG-mapping procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Golda Nicholas, MD, Principal Investigator — 573-882-8578
Locations (1):
- University of Missouri Health Care, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided